CLINICAL TRIAL: NCT04136470
Title: Development of BioForte Technology for in Silico Identification of Valuable Genomic Features That Are Candidates for Microbiome-based Therapeutics and Diagnostics.
Brief Title: BioForte Technology for in Silico Identification of Candidates for a New Microbiome-based Therapeutics and Diagnostics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ardigen (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: BioForte; POIR.01.01.01-00-0347/17 (Other Grant/Funding Number: The National Centre for Research and Development)
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Non Small Cell Lung Cancer; Microbiome; Metagenome; Immunotherapy; Melanoma
Keywords: Microbiome; Cancer; Metagenome; Non Small Cell Lung Cancer; Immunotherapy; Neoplasms; Nivolumab; Ipilimumab; Atezolizumab; Stool; FFPE; PBMC; Intestinal microbiota; Immuno-Oncology; Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Neoplasms | interventions — Blood Specimen Collection; Biopsy; Nivolumab; Ipilimumab; atezolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — stool, biopsy (FFPE) and peripheral blood samples (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC: This cohort will consist of 100 patients with non-small cell lung cancer (NSCLC).
  Interventions: Biological: Collection of stool, blood (PBMC) and biopsy (FFPE)
- MEL: This cohort will consist of 30 patients with melanoma (MEL).
  Interventions: Biological: Collection of stool, blood (PBMC) and biopsy (FFPE)

INTERVENTIONS:
Biological: Collection of stool, blood (PBMC) and biopsy (FFPE) — Patients receiving routine treatment (immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies), financed by the Polish National Health Fund (NFZ).
  Other Names: Nivolumab; Ipilimumab; Atezolizumab

SUMMARY:
The goal of the project is to develop and validate the BioForte technology. Its main functionality should be to in silico determine candidates for novel microbiome-based therapeutics and diagnostics. Key challenge to be solved using the technology is to detect the differences in gut microbiome between oncology patients who respond to immunotherapies and the ones who do not respond to this treatment.

This technology employs machine learning methods to replace the laboratory procedure for finding valuable genomic features. Such features can be crucial to identify differences between the two populations (e.g. responders vs non-responders) to target specific strains.

The samples and data collected in this clinical study will be used for clinical validation of BioForte technology. For all patients treated with immunotherapy, stool collection will be performed per patient (one stool collection before setting up immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies). Samples will be sequenced by long-read sequencing technology. In parallel, we will also collect samples of peripheral blood samples (PBMC) and biopsy (FFPE).

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age.
* Patients with one of the following types of cancer: non-small cell lung cancer, melanoma.
* Patients with informed consent to participate in the study.
* Patients receiving routine treatment (immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies), financed by the Polish National Health Fund (NFZ).
* The applied immunotherapy should be the first or second line of treatment.

Exclusion Criteria:

* Patients who are unable to understand, read and / or sign informed consent.
* Patients who can not collect stools.
* Patients with fecal transplant.
* The applied immunotherapy is not the first or second line of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving routine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Microbial diversity in stool samples | Inclusion
  Microbila DNA - stool samples sequenced by long-read sequencing technology.
Number of Responders and Non-responders on immunotherapy (evaluated using RECIST 1.1 criteria) | Up to 6 months
  Standard follow-up care after cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Warchol, PhD, Principal Investigator — Ardigen
Locations (10):
- Poland (10):
  - University Clinical Centre in Gdansk, Gdansk
  - The John Paul II Hospital in Krakow, Krakow
  - The Maria Sklodowska-Curie National Research Institute of Oncology Krakow Branch, Krakow
  - Poznań University Hospital of Lord's Transfiguration, Poznan
  - Provincial Hospital St. Father Pio in Przemyśl, Przemyśl
  - Mountains Center of Pulmonology and Chemotherapy "Izer-Med", Szklarska Poręba
  - Specialist Oncological Hospital, Tomaszów Mazowiecki
  - The Maria Sklodowska-Curie National Research Institute of Oncology in Warsaw, Warsaw
  - Masovian Oncology Hospital in Wieliszew, Wieliszew
  - Lower Silesian Oncology Center & Łukasiewicz Research Network - PORT Polish Center For Technology Development, Wroclaw